CLINICAL TRIAL: NCT02818998
Title: An Open-label, Randomized, Active-controlled, Parallel-group, Phase-3b Study of the Efficacy, Safety, and Tolerability of Three Different Treatment Regimens of 2 mg Aflibercept Administered by Intravitreal Injections to Subjects With Diabetic Macular Edema (DME)
Brief Title: Efficacy and Safety of Three Different Aflibercept Regimens in Subjects With Diabetic Macular Edema (DME)
Acronym: VIOLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17613; 2014-004938-25 (EudraCT Number)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Macular Edema
Keywords: Diabetic macular edema; DME
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aflibercept 2 mg fixed (Experimental): Participants received fixed dosing of 2 mg aflibercept at injection intervals of 8 weeks
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Aflibercept 2 mg flexible (Experimental): Participants received flexible dosing of 2 mg aflibercept at injection intervals of ≥8 week
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Aflibercept 2 mg PRN (Experimental): Participants received monthly monitoring with 2 mg aflibercept injection pro re nata (PRN, as needed)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

SUMMARY:
To evaluate the efficacy of long-term treatment with 2 mg aflibercept via different intravitreal (IVT) treatment regimens to participants with DME pretreated with 2 mg aflibercept every 8 weeks after 5 initial monthly injections for approximately 1 year or more (according to the EU label for the first year of treatment)

ELIGIBILITY:
Inclusion Criteria:

The subject's history of aflibercept treatment met all of the following:

* Treatment in the study eye was initiated with five monthly (-1 week /+2 weeks) doses of 2 mg aflibercept and improvements of visual and anatomic outcomes were observed and documented.
* Following the above initiation phase, the intervals between treatments were between 6 weeks and 12 weeks (one exception was allowed).
* The interval between the last 2 pre-study injections was ≥ 8 weeks, and visual and anatomic outcomes had been stable over this interval.
* The subject received the last intravitreal (IVT) injection of aflibercept in the study eye 8 weeks (±10 days) before the first planned treatment /randomization in this study.
* Total prior treatment duration with aflibercept (i.e. from first aflibercept treatment ever to enrollment into this study) was 1 year or longer.

To be met at initiation of pre-study aflibercept treatment:

* Type 1 or 2 diabetes mellitus (DM)
* Diagnosis of diabetic macular edema (DME) secondary to DM involving the center of the macula (defined as the area of the center subfield on optical coherence tomography [OCT]) in the study eye
* Decrease in vision determined to be primarily the result of DME in the study eye
* Best corrected visual acuity (BCVA) in the study eye of Early Treatment Diabetic Retinopathy Study (ETDRS) letter score 73 to 24

Exclusion Criteria:

At initiation of pre-study aflibercept treatment:

- Previous treatment with anti-angiogenic drugs in study eye (e.g., pegaptanib sodium, bevacizumab, ranibizumab, or aflibercept) within the last 12 weeks before initiation of aflibercept pre-study treatment

At initiation of pre-study aflibercept treatment, screening for this study, and baseline for this study:

* Prior treatment of the study eye with long acting steroids, either periocular or intraocular, in the preceding 120 days or Iluvien intravitreal implant at any time
* Active proliferative diabetic retinopathy, current iris neovascularization, vitreous hemorrhage, or tractional retinal detachment in the study eye
* Cataract surgery or any other intraocular surgery within 90 days of aflibercept treatment in the study eye
* Ocular inflammation (including trace or above) or history of uveitis in the study eye
* Structural damage to the center of the macula in the study eye that was likely to preclude improvement in BCVA following the resolution of macular edema including atrophy of the retinal pigment epithelium, subretinal fibrosis or scar, significant macular ischemia or organized hard exudates
* Concurrent disease in the study eye, other than DME, that could compromise visual acuity, require medical or surgical intervention during the study period, or could confound interpretation of the results (including advanced glaucoma, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause)
* Uncontrolled DM as defined by hemoglobin (Hb) A1c > 12.0% at screening and baseline for this study
* Any ocular or periocular infection in the preceding 4 weeks in either eye
* History of either cerebral vascular accident and/or myocardial infarction within 180 days before aflibercept treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (58):
- Austria (2):
  - Graz, Styria
  - Vienna
- Canada (5):
  - Halifax, Nova Scotia
  - Mississauga, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Czechia (2):
  - Hradec Králové
  - Prague
- Créteil, France
- Germany (7):
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dresden, Saxony
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Italy (8):
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Florence, Tuscany
  - Padua, Veneto
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (8):
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
- Portugal (5):
  - Vila Franca de Xira, Lisbon District
  - Coimbra
  - Leiria
  - Lisbon
  - Porto
- Slovakia (4):
  - Bratislava
  - Nitra
  - Zvolen
  - Žilina
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - Sant Cugat Del Vallés, Barcelona
  - Albacete
  - Barcelona
  - Valencia
- Switzerland (2):
  - Bern
  - Geneva
- United Kingdom (4):
  - Southampton, Hampshire
  - Sunderland, Tyne and Wear
  - Leeds, West Yorkshire
  - London

REFERENCES:
- [Derived] Garweg JG, Stefanickova J, Hoyng C, Niesen T, Schmelter T, Leal S, Sivaprasad S; VIOLET Investigators. Dosing Regimens of Intravitreal Aflibercept for Diabetic Macular Edema Beyond the First Year: VIOLET, a Prospective Randomized Trial. Adv Ther. 2022 Jun;39(6):2701-2716. doi: 10.1007/s12325-022-02119-z. Epub 2022 Apr 12. PMID 35412227
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 14 countries between 16-Nov-2016 (first participant first visit) and 24-Sep-2019 (last participant last visit).
Pre-assignment Details: A total of 500 participants were screened in this study. Of these, 37 participants did not enter the treatment period (31 were screening failures; 3 were lost to follow-up; 2 had an adverse event (AE) and 1 was not randomized due to an "other" reason). A total of 463 participants were randomized and received treatment.
Groups:
- Aflibercept 2 mg Extended: Participants received flexible dosing of 2 mg aflibercept at injection intervals of ≥8 weeks
Period: Overall Study
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Started | 155 | 154 | 154
Completed Week 52 Visit | 144 | 146 | 140
Completed (Completed Week 100 visit) | 137 | 138 | 136
Not Completed | 18 | 16 | 18
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Lost to Follow-up | 4 | 1 | 2
Not completed — Withdrawal by sponsor | 0 | 1 | 1
Not completed — Death | 3 | 6 | 8
Not completed — Withdrawal by Subject | 7 | 6 | 6
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): included all participants who received any study drug under the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN | Total
Number analyzed (Participants) | 155 | 154 | 154 | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.7) | 64.8 (10.1) | 65.4 (9.3) | 64.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 59 | 64 | 178
  Male | 100 | 95 | 90 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 7
  Not Hispanic or Latino | 144 | 142 | 142 | 428
  Unknown or Not Reported | 10 | 10 | 8 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 141 | 144 | 147 | 432
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 7 | 27
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: Scores on a scale] — Best Corrected Visual Acuity (BCVA) was measured in the study eye by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. The ETDRS chart includes 70 letters in total and the letter score ranges from 0 to 100. More letters read correctly results in a higher letter score, which represents better visual acuity.
  Scores on a scale | 72.8 (10.38) | 72.5 (11.35) | 71.0 (10.87) | 72.1 (10.88)
Central Retinal Thickness (CRT) [Mean (Standard Deviation); unit: Microns] — Central Retinal Thickness (CRT) was measured in the study eye by spectral domain optical coherence tomography (SD-OCT).
  Microns | 289.8 (66.46) | 285.3 (76.01) | 294.5 (80.72) | 289.9 (74.55)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 52
Description: Best Corrected Visual Acuity (BCVA) was measured in the study eye by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. The ETDRS chart includes 70 letters in total and the letter score ranges from 0 to 100. More letters read correctly results in a higher letter score, which represents better visual acuity.
Time Frame: From baseline to Week 52
Population: Full Analysis Set (FAS): included all randomized participants who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 153 | 152 | 153
Scores on a scale | 0.4 (6.7) | 0.5 (6.7) | 1.7 (6.8)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Non-Inferiority — Non-inferiority margin: 4 letters; p < 0.0001, ANCOVA — Non-inferiority was demonstrated if the p-value (adjusted for multiplicity using the Hochberg procedure) was < 0.025; Least Squares mean difference = 0.01, 95% CI 2-sided [-1.46 to 1.47]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Non-Inferiority — Non-inferiority margin: 4 letters; p < 0.0001, ANCOVA — Non-inferiority was demonstrated if the p-value (adjusted for multiplicity using the Hochberg procedure) was < 0.025; Least Squares mean difference = 0.95, 95% CI 2-sided [-0.52 to 2.42]

2. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) at Week 52
Description: Central Retinal Thickness (CRT) was measured in the study eye by spectral domain optical coherence tomography (SD-OCT).
Time Frame: From baseline to week 52
Population: Participants in FAS taken into account for this analysis
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 147 | 147 | 153
Microns | -18.8 (45.5) | -2.1 (56.2) | 2.2 (77.8)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; p = 0.0105, ANCOVA; Least Square mean difference = 14.38, 95% CI 2-sided [3.39 to 25.37]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; p = 0.0023, ANCOVA; Least Square mean difference = 21.22, 95% CI 2-sided [7.65 to 34.80]

3. Secondary Outcome: Number of Participants With Categorized Changes From Baseline in Best Corrected Visual Acuity (BCVA) at Week 52
Description: as for outcome 1
Time Frame: From baseline to week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 153 | 152 | 153
Participants
  ≥15 letter gain | 4 | 5 | 4
  ≥10 letter gain | 10 | 14 | 13
  ≥30 letter loss | 1 | 0 | 0
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥ 15 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 0.68, 95% CI 2-sided [-3.14 to 4.49]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥10 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 2.66, 95% CI 2-sided [-3.40 to 8.73]
Statistical Analysis 3: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥30 letter loss: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = -0.66, 95% CI 2-sided [-1.94 to 0.63]
Statistical Analysis 4: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥15 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = -0.13, 95% CI 2-sided [-3.68 to 3.41]
Statistical Analysis 5: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥10 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 1.72, 95% CI 2-sided [-4.10 to 7.54]
Statistical Analysis 6: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥30 letter loss: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = -0.68, 95% CI 2-sided [-2.00 to 0.65]

4. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 100
Description: as for outcome 1
Time Frame: From baseline to Week 100
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 153 | 152 | 153
Scores on a scale | 0.1 (7.2) | -0.1 (9.1) | 1.8 (9.0)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Non-Inferiority — Non-inferiority margin: 4 letters; p < 0.0001, ANCOVA; Least Squares mean difference = -0.30, 95% CI 2-sided [-2.13 to 1.52]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Non-Inferiority — Non-inferiority margin: 4 letters; p < 0.0001, ANCOVA; Least Squares mean difference = 1.39, 95% CI 2-sided [-0.40 to 3.19]

5. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) at Week 100
Description: Central Retinal Thickness (CRT) was measured in the study eye by spectral domain optical coherence tomography (SD-OCT).
Time Frame: From baseline to Week 100
Population: Participants in FAS taken into account for this analysis
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 147 | 147 | 153
Microns | -15.5 (64.3) | 2.3 (81.8) | -13.9 (74.4)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; p = 0.0416, ANCOVA; Least Square mean difference = 16.14, 95% CI 2-sided [0.62 to 31.66]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; p = 0.5524, ANCOVA; Least Square mean difference = 4.12, 95% CI 2-sided [-9.52 to 17.77]

6. Secondary Outcome: Number of Participants With Categorized Changes From Baseline in Best Corrected Visual Acuity (BCVA) at Week 100
Description: as for outcome 1
Time Frame: From baseline to Week 100
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 153 | 152 | 153
Participants
  ≥15 letter gain | 3 | 4 | 6
  ≥10 letter gain | 10 | 17 | 22
  ≥30 letter loss | 1 | 2 | 2
Statistical Analysis 1: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥ 15 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 0.67, 95% CI 2-sided [-2.72 to 4.05]
Statistical Analysis 2: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥10 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 4.63, 95% CI 2-sided [-1.73 to 10.98]
Statistical Analysis 3: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg Extended; ≥30 letter loss: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 0.66, 95% CI 2-sided [-1.56 to 2.87]
Statistical Analysis 4: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥15 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 1.90, 95% CI 2-sided [-1.89 to 5.69]
Statistical Analysis 5: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥10 letter gain: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 7.54, 95% CI 2-sided [0.81 to 14.28]
Statistical Analysis 6: Comparison: Aflibercept 2 mg Fixed vs Aflibercept 2 mg PRN; ≥30 letter loss: Aflibercept 2 mg fixed was regarded as the reference arm; Test type: Other; Cochran-Mantel-Haenszel; Treatment Difference = 0.63, 95% CI 2-sided [-1.61 to 2.88]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAE)
Description: AEs that started after the first application of aflibercept under this protocol until 30 days after the last dose of study drug administration
Time Frame: Up to Week 100
Population: Safety analysis set (SAF): included all participants who received any study drug under the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
Number analyzed (Participants) | 155 | 154 | 154
Participants | 129 | 128 | 129

ADVERSE EVENTS:
Time Frame: After the first application of Aflibercept under this protocol and within 30 days after the last dose of study drug administration, assessed up to Week 100.
Groups:
- Aflibercept 2 mg Extended: Participants received flexible dosing of 2 mg aflibercept at injection intervals of >=8 week
Arm/Group | Aflibercept 2 mg Fixed | Aflibercept 2 mg Extended | Aflibercept 2 mg PRN
All-Cause Mortality (participants affected / at risk) | 3/155 | 6/154 | 8/154
Serious Adverse Events (participants affected / at risk) | 35/155 | 38/154 | 37/154
Other Adverse Events (participants affected / at risk) | 97/155 | 85/154 | 98/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Fixed (N=155) | Aflibercept 2 mg Extended (N=154) | Aflibercept 2 mg PRN (N=154)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (4) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign spleen tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Heart valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 2 (2) | 1 (1) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Fixed (N=155) | Aflibercept 2 mg Extended (N=154) | Aflibercept 2 mg PRN (N=154)
Cataract (Eye disorders) | 27 (37) | 29 (41) | 24 (35)
Cataract cortical (Eye disorders) | 8 (11) | 7 (10) | 6 (10)
Cataract nuclear (Eye disorders) | 9 (11) | 0 (0) | 7 (8)
Cataract subcapsular (Eye disorders) | 7 (10) | 9 (10) | 8 (10)
Diabetic retinal oedema (Eye disorders) | 12 (15) | 13 (17) | 14 (17)
Diabetic retinopathy (Eye disorders) | 14 (18) | 14 (18) | 18 (23)
Macular oedema (Eye disorders) | 8 (10) | 11 (14) | 17 (32)
Maculopathy (Eye disorders) | 3 (4) | 1 (2) | 13 (20)
Posterior capsule opacification (Eye disorders) | 5 (6) | 9 (9) | 10 (12)
Retinal haemorrhage (Eye disorders) | 4 (7) | 3 (3) | 10 (21)
Visual acuity reduced (Eye disorders) | 25 (42) | 22 (30) | 22 (30)
Cystoid macular oedema (Eye disorders) | 14 (25) | 12 (17) | 10 (15)
Macular fibrosis (Eye disorders) | 7 (7) | 6 (7) | 10 (11)
Conjunctivitis (Infections and infestations) | 4 (7) | 1 (1) | 8 (12)
Influenza (Infections and infestations) | 8 (8) | 3 (3) | 8 (8)
Nasopharyngitis (Infections and infestations) | 14 (18) | 14 (18) | 17 (24)
Intraocular pressure increased (Investigations) | 11 (14) | 4 (5) | 11 (14)
Diabetes mellitus (Metabolism and nutrition disorders) | 24 (26) | 10 (10) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT02818998/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02818998/SAP_001.pdf